CLINICAL TRIAL: NCT03202888
Title: Novel IT to Create Patient-Integrated Hospital Quality Improvement and Improve Patient Safety
Brief Title: Family Input for Quality and Safety
Acronym: FIQS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FIQS
Record Dates: First submitted 2017-06-20; First posted 2017-06-29 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Patient Safety
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): After completing enrollment surveys, including measures of patient activation and medical knowledge, participants will be invited to use the novel IT. The technology is a mobile responsive website for survey data collection made by our technology vendor, QuesGen. Patients and family members will be able to access the website from any personal device with internet access: laptop, tablet, or smart phone. QuesGen will send a text message reminder to participants with a link to specific questionnaires at scheduled time intervals. Frequency of text messaging will likely be daily, but will ultimately reflect family and patient feedback in Aim 1. In addition to text reminders, participants will be able to answer questionnaires at-will by accessing the mobile responsive website.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — QuesGen-created mobile responsive website tool, Family Input for Quality and Safety.

SUMMARY:
This project aims to create and evaluate a tool that gathers patient and family member feedback and makes it rapidly available to providers, enabling nimble and responsive safety and quality improvement efforts. Aim 1. Determine feasibility and acceptability of the patient data collection and provider dashboard tool. The investigators will conduct usability testing prior to study start, measure user (patients and providers) engagement over time, and gather feedback about the tool at study end. This will test the hypothesis that patient and caregiver characteristics will predict tool use. Aim 2. Assess whether reporting patient- and caregiver- observed processes of care to providers leads to changes over time. The investigators hypothesize that performance on structured items of interest will improve over time with rapidly available data presented to providers. Aim 3. Estimate tool implementation effect sizes, using a pre-post design, on medical errors.

DETAILED DESCRIPTION:
More than a decade after the seminal Institute Of Medicine report, "To Err is Human", failure rates in patient safety remain stubbornly high in hospitals. Prior efforts to improve hospital quality have had relatively little impact, in part due to limited access to timely quality improvement data. The long-term goal of this application is to leverage existing technologies to give voice to hospitalized patients and their family members, leading to improvements in hospital safety and quality. The overall objective in this application is to create and evaluate a tool that gathers patient and family member feedback and makes it rapidly available to providers, enabling nimble and responsive safety and quality improvement efforts. The central hypothesis, based on the theory of co-production, is that observations from patients and families, gathered in a structured way, will provide actionable information regarding patient safety and quality. The rationale for doing this project is to test an innovative new approach to creating a rapidly available data stream to providers who are working on specific improvement efforts, and a mechanism for creating a quality improvement approach that is inherently patient-centered. The investigators plan to test the central hypothesis and thereby accomplish the objective of this application by focusing on the following areas of research for Health IT: Use, Implementation, and Impact on Outcomes, under the study type "Pilot and feasibility", pursuing three specific aims: Aim 1. Determine feasibility and acceptability of the patient data collection and provider dashboard tool (Use and Implementation). The investigators will conduct usability testing prior to study start, measure user (patients and providers) engagement over time, and gather feedback about the tool at study end. The investigators hypothesize that patient and caregiver characteristics will predict tool use. Aim 2. Assess whether reporting patient- and caregiver- observed processes of care to providers leads to changes over time (Implementation). The investigators hypothesize that performance on structured items of interest will improve over time with rapidly available data presented to providers. Aim 3. Estimate tool implementation effect sizes, using a pre-post design, on medical errors (Impact on outcomes). The proposed research is innovative, in the investigators' opinion, based on a paradigm-shifting conceptual model of patient-engaged quality improvement, and because it leverages technology to gather and present data in an unprecedented manner. The expected contribution of the proposed research will be an adapted tool that will gather meaningful and important data on patient safety and present it in an actionable way to providers and hospital leaders, resulting in a powerful data stream to fuel rapid improvements in patient safety. Pilot data from this proposal will inform the design of a future cluster-randomized trial of the new tool across multiple hospital systems. This contribution will be significant because it represents key steps towards a new approach to improving patient safety in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient and caregiver participants will be recruited from admitted patients and their family members on the medical-surgical units at UCSF's Benioff Children's Hospital during the study period.
* Eligible providers will be the participating hospitalists during the study period.

All nurse managers on the units and the patient safety and quality managers for the units will be eligible. All nurses will be eligible on the participating units.

Exclusion Criteria:

* Patients who are youth in the foster care system will not be eligible.
* Patients or parents/guardians who do not have smart phones will not be eligible.

There are no provider or nurse or quality manager exclusions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Change in rate of preventable medical errors or adverse events per 100 admissions | Measured cross-sectionally in the hospital unit at baseline for three months, and again for three months at the end of the intervention (months 10,11,12 of the intervention).
  This is a hospital unit-level outcome measure, assessing unit-level rate of adverse events and preventable medical errors in a time period before the intervention, and the unit-level rate at the end of the intervention. The investigators will apply standard definitions of medical errors as preventable failures in processes of care and adverse events as preventable and non-preventable unintended consequences of medical care that lead to patient harm. This is a composite measure and will be measured as total count of medical errors plus total count of adverse events per 100 admissions. The investigators will not track this measure across the same group of patients in the before and after periods. Participants will be included for the duration of their admission, which may vary. The rate will be measured cross-sectionally in both time periods.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Bardach, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James JT. A new, evidence-based estimate of patient harms associated with hospital care. J Patient Saf. 2013 Sep;9(3):122-8. doi: 10.1097/PTS.0b013e3182948a69. PMID 23860193
- [Background] Classen DC, Resar R, Griffin F, Federico F, Frankel T, Kimmel N, Whittington JC, Frankel A, Seger A, James BC. 'Global trigger tool' shows that adverse events in hospitals may be ten times greater than previously measured. Health Aff (Millwood). 2011 Apr;30(4):581-9. doi: 10.1377/hlthaff.2011.0190. PMID 21471476
- [Background] Shekelle PG, Pronovost PJ, Wachter RM, Taylor SL, Dy SM, Foy R, Hempel S, McDonald KM, Ovretveit J, Rubenstein LV, Adams AS, Angood PB, Bates DW, Bickman L, Carayon P, Donaldson L, Duan N, Farley DO, Greenhalgh T, Haughom J, Lake ET, Lilford R, Lohr KN, Meyer GS, Miller MR, Neuhauser DV, Ryan G, Saint S, Shojania KG, Shortell SM, Stevens DP, Walshe K. Advancing the science of patient safety. Ann Intern Med. 2011 May 17;154(10):693-6. doi: 10.7326/0003-4819-154-10-201105170-00011. PMID 21576538
- [Background] Landrigan CP, Parry GJ, Bones CB, Hackbarth AD, Goldmann DA, Sharek PJ. Temporal trends in rates of patient harm resulting from medical care. N Engl J Med. 2010 Nov 25;363(22):2124-34. doi: 10.1056/NEJMsa1004404. PMID 21105794
- [Background] Chassin MR. Improving the quality of health care: what's taking so long? Health Aff (Millwood). 2013 Oct;32(10):1761-5. doi: 10.1377/hlthaff.2013.0809. PMID 24101066
- [Background] Erasmus V, Daha TJ, Brug H, Richardus JH, Behrendt MD, Vos MC, van Beeck EF. Systematic review of studies on compliance with hand hygiene guidelines in hospital care. Infect Control Hosp Epidemiol. 2010 Mar;31(3):283-94. doi: 10.1086/650451. PMID 20088678
- [Background] Conway PH, Mostashari F, Clancy C. The future of quality measurement for improvement and accountability. JAMA. 2013 Jun 5;309(21):2215-6. doi: 10.1001/jama.2013.4929. No abstract available. PMID 23736730
- [Background] Blumenthal D, McGinnis JM. Measuring Vital Signs: an IOM report on core metrics for health and health care progress. JAMA. 2015 May 19;313(19):1901-2. doi: 10.1001/jama.2015.4862. No abstract available. PMID 25919301
- [Background] Rossi P, Lipsey M, Freeman H. Evaluation: A Systematic Approach. 7th Edition ed: SAGE Publications, Inc; 2003.
- [Background] Bardach NS, Asteria-Penaloza R, Boscardin WJ, Dudley RA. The relationship between commercial website ratings and traditional hospital performance measures in the USA. BMJ Qual Saf. 2013 Mar;22(3):194-202. doi: 10.1136/bmjqs-2012-001360. Epub 2012 Nov 23. PMID 23178860
- [Background] Greaves F, Pape UJ, King D, Darzi A, Majeed A, Wachter RM, Millett C. Associations between Web-based patient ratings and objective measures of hospital quality. Arch Intern Med. 2012 Mar 12;172(5):435-6. doi: 10.1001/archinternmed.2011.1675. Epub 2012 Feb 13. No abstract available. PMID 22331980
- [Background] Greaves F, Pape UJ, King D, Darzi A, Majeed A, Wachter RM, Millett C. Associations between Internet-based patient ratings and conventional surveys of patient experience in the English NHS: an observational study. BMJ Qual Saf. 2012 Jul;21(7):600-5. doi: 10.1136/bmjqs-2012-000906. Epub 2012 Apr 20. PMID 22523318
- [Background] Han E, Hudson Scholle S, Morton S, Bechtel C, Kessler R. Survey shows that fewer than a third of patient-centered medical home practices engage patients in quality improvement. Health Aff (Millwood). 2013 Feb;32(2):368-75. doi: 10.1377/hlthaff.2012.1183. PMID 23381530
- [Background] Clancy CM. Where we are a decade after To err is human. J Patient Saf. 2009 Dec;5(4):199-200. doi: 10.1097/PTS.0b013e3181c2114a. No abstract available. PMID 22130210
- [Background] Guide to Patient and Family Engagement: Environmental Scan Report. October 2014; http://www.ahrq.gov/research/findings/final-reports/ptfamilyscan/ptfamilysum.html. Accessed June 10, 2015.